CLINICAL TRIAL: NCT06826859
Title: Dose Based Aspirin Pharmacokinetics and Pharmacodynamics in Pregnancy and Association With Pregnancy Outcomes
Brief Title: Daily Aspirin vs Split Dosing in High-risk Pregnancies (DASH)
Acronym: DASH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRISID-2024-1554; 1R01HD112076 (NIH)
Record Dates: First submitted 2025-01-28; First posted 2025-02-14 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Preterm Birth; Preeclampsia
Keywords: Aspirin; Preeclampsia; Preterm birth; Pregnancy; Pharmacokinetics; Pharmacodynamics; Phase I/II; Randomized clinical trial
MeSH Terms: conditions — Premature Birth; Pre-Eclampsia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Biostatistical analysis, all laboratory assessments will be conducted by personnel blinded to study groupl
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Daily aspirin (Active Comparator): 162mg aspirin daily
  Interventions: Drug: Daily aspirin (ASA)
- Split dose aspirin (Experimental): 81mg aspirin q12 hours
  Interventions: Drug: Split dose aspirin (ASA)

INTERVENTIONS:
Drug: Daily aspirin (ASA) — 162mg aspirin taken daily
  Arms: Daily aspirin
Drug: Split dose aspirin (ASA) — 81mg aspirin q12hours
  Arms: Split dose aspirin

SUMMARY:
Aspirin is recommended in high risk patients to reduce the risk of preeclampsia and preterm birth, which are leading causes of both maternal and neonatal morbidity and mortality, but up to 20% will have these adverse outcomes despite therapy. Gaps in knowledge regarding pregnancy specific aspirin pharmacology and the relationship of aspirin response and pregnancy outcome, along with a lack of consensus on aspirin dosing has limited the effective use of this intervention. The investigators aim to apply principles of clinical pharmacology to determine how to optimally utilize this low cost medication to improve maternal/child health outcomes. This is a Phase I/II randomized controlled trial of high risk pregnancies recommended aspirin; participants will be randomized to take aspirin either 162mg once daily, or 81mg twice a day. Outcomes evaluated will include the difference in aspirin response between these two dosing regimens, the individual factors that impact aspirin pharmacology in pregnancy, and evaluate markers or aspirin response that may be associated with pregnancy outcome.

DETAILED DESCRIPTION:
This is an unblinded randomized controlled Phase I/II trial comparing high risk singleton pregnancies randomized to 162mg daily (daily dose) vs 81mg q12hours (split dose). Participants will be enrolled prior to 16 weeks gestation. The primary outcome is platelet inhibition as assessed by PFA-100 epinephrine closure time, assessed 2-4 weeks after initiation and again at 28-32 weeks gestation. A subset of participants will be enrolled in a pharmacokinetic study to evaluate pharmacokinetics of aspirin in pregnancy at the two dosing intervals. Secondary outcomes include urine thromboxane at each visit, platelet associated microRNAs. Individual factors associated with aspirin pharmacokinetics and pharmacodynamics in pregnancy will be assessed. Finally, the relationship between these pharmacodynamic markers and pregnancy outcome will be evaluated.

ELIGIBILITY:
Inclusion Criteria

* Singleton gestation gestational age <16 0/7 weeks, dating confirmed with ultrasound
* ≥1 high risk factor for preeclampsia or ≥2 moderate risk factors as per United States Preventative Services Task Force (2021)
* Recommendation for 162mg aspirin daily in pregnancy
* Age 16-55 years old

Exclusion criteria

* Contraindication to aspirin
* Current or planned use of any other anticoagulation
* Thrombocytopenia, other known platelet or bleeding disorder
* Abnormally elevated baseline PFA-100 epinephrine closure time prior to aspirin initiation

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-06-26 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Aspirin Response PFA-100 epinephrine closure time (seconds) | 2-4 weeks after aspirin initiation
  Difference in PFA-100 epinephrine closure time (seconds)

SECONDARY OUTCOMES:
Aspirin response (PFA-100 epinephrine closure time) | 28-32 weeks gestation
  Difference in PFA-100 epinephrine closure time (seconds)
Urinary thromboxane concentration | 2-4 weeks after aspirin initiation
  Difference in Urine thromboxane (AspirinWorks)
Urinary Thromboxane concentration | 28-32 weeks gestation
  Difference in Urinary thromboxane (AspirinWorks)
Inadequate aspirin response | 2-4 weeks after aspirin initiation
  Number of participants with PFA-100 epinephrine closure time<150 seconds
Inadequate aspirin response | 28-32 weeks gestation
  Number of participants with PFA-100 epinephrine closure time<150seconds
Preterm birth | Delivery
  Number of participants with Preterm birth<37 weeks
Indicated preterm birth | delivery
  Number of participants with Preterm birth<37 weeks due to preeclampsia or fetal growth restriction
Spontaneous preterm birth | delivery
  Number of participants with spontaneous preterm birth <37 weeks
MicroRNAs | 2-4 weeks after aspirin initiation
  Fold-change from baseline for concentration of circulating microRNAs
MicroRNAs | 28-32 weeks gestation
  Fold-change from baseline for concentration of circulating microRNAs
Placental histopathology | Delivery
  Placental pathology per Amsterdam criteria. Number of participants with maternal vascular malperfusion, intervillous thrombosis
Birthweight | Delivery
  Infant birthweight (grams)
Fetal growth restriction | delivery
  Number of participants diagnosed with Fetal growth restriction
Hypertensive disorder of pregnancy | delivery
  Number of participants diagnosed with Preeclampsia or gestational hypertension
Gestational age at delivery | Delivery
  Gestational age at delivery (weeks)
Pregnancy loss<20 weeks | delivery
  Number of participants with Pregnancy loss (delivery, demise, miscarriage)<20 weeks gestation
Fetal demise | delivery
  Number of participants with Fetal demise diagnosed >=20 weeks gestation
Antepartum bleeding | Delivery
  Number of participants with any admission for antepartum bleeding
Abruption | delivery
  Number of participants with Abruption diagnosed prior to or at delivery
Placental hematoma | delivery
  Number of participants with Placental hematoma suspected on ultrasound
Postpartum hemorrhage | Delivery
  Number of participants with Postpartum hemorrhage >1000ml
Adherence | 2-4 weeks after aspirin
  Number of participants with Adherence>75%
Adherence | 28-32 weeks
  Number of participants with Adherence>75%
Neonatal intraventricular hemorrhage Grade II or higher | Neonatal discharge
  Number of participants with infants found to have Neonatal IVH grade II or higher diagnosed on ultrasound post natally
Cordblood serum thromboxane | Delivery
  cordblood serum thromboxane concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be submitted to NICHD DASH and can be requested through NICHD DASH
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 1 year after study completion
Access Criteria: Data will be submitted to NICHD DASH and may be requested through DASH
URL: https://dash.nichd.nih.gov/